CLINICAL TRIAL: NCT06474715
Title: Cluster Randomized Controlled Trial to Promote Physical Activity Among Low-resourced Mothers in New York City: Protocol for the Free Time for Wellness (FT4W) Effectiveness Trial.
Brief Title: Free Time For Wellness Pilot Effectiveness Trial
Acronym: FT4W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Monash University (Other); Loughborough University (Other); University of Iowa (Other); Public Health Institute (Unknown); Jovie USA, LLC (Industry); West Side Campaign Against Hunger (Unknown); New York City Parks and Recreation (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lauren C. Houghton, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAU8303 - Pilot; 5R01MD018609 (NIH)
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Physical Inactivity
Keywords: Motherhood; Childcare; Social cohesion
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The FT4W program is founded on social cognitive theory, which posits that human behavior is the product of the dynamic interplay of personal, behavioral, and environmental influences. Social cognitive theory emphasizes reciprocal determinism in interactions between people and their environments. The majority of physical activity interventions use social cognitive theory as indicated by the theory and technique tool developed by the Human Behavior Change Project. The study team also used the theory and technique tool to align the FT4W program components and mediating pathways with behavior change techniques and mechanisms of action substantiated in behavior change literature and expert consensus. For our study, the study team will measure social influence via social cohesion.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm: Fitness classes only (No Intervention): There will be 3 Shape Up NYC classes offered weekly for one hour free of charge to consenting participants in all three arms with a total of 12 classes offered per participant.
  Weekly reminders for each class will be sent via automated text messages to individuals.
- Comparator Arm: Fitness classes + childcare (Active Comparator): There will be 3 Shape Up NYC classes offered weekly for one hour free of charge to consenting participants in all three arms with a total of 12 classes offered per participant.
  In addition, they will receive childcare in an adjacent space to the fitness class.
  Weekly reminders for each class will be sent via automated text messages to individuals.
  Interventions: Behavioral: Arms
- Enhanced intervention arm: Fitness classes + childcare + peer support (Experimental): There will be 3 Shape Up NYC classes offered weekly for one hour free of charge to consenting participants in all three arms with a total of 12 classes offered per participant.
  In addition, they will receive childcare in an adjacent space to the fitness class.
  In addition to childcare, Arm C will also receive peer support activities. Peer support activities will consist of group volunteer activities at food pantries, free deliveries of food pantry groceries, and group play dates at local playgrounds. A Community Champion will also facilitate group text messages.
  Interventions: Behavioral: Arms

INTERVENTIONS:
Behavioral: Arms — The intervention includes a task-based interaction (volunteer activities) where cognitive demand is low and interactional roles are clear. The focus is on the task, rather than developing relationships, reducing the pressure of interaction. As the volunteer activities continue, they also offer the opportunity for group members to enhance empathy, another salient component of cross-group relational development. Mediated interaction supports new relational development through a disinhibiting effect, lowering inhibitions and increasing comfort and disclosure
  Arms: Comparator Arm: Fitness classes + childcare; Enhanced intervention arm: Fitness classes + childcare + peer support

SUMMARY:
Physical inactivity is pervasive and prevalent in the United States, particularly among women of low socioeconomic position, and women with children. Structural and social barriers make active leisure time a rare commodity creating a pressing health issue because physical inactivity increases the risk of chronic diseases and poor health. The broad objective of this study is to pilot test the Free Time for Wellness (FT4W), an innovative multilevel physical activity intervention to increase physical activity among low-resourced mothers.

DETAILED DESCRIPTION:
Physical inactivity is particularly prevalent in women of low socioeconomic position (SEP) (60% are inactive), suggesting that there are structural barriers to being physically active. This study will pilot test the intervention to increase physical activity among mothers of low SEP, where there is high risk of chronic disease and significant potential to make an impact on these health disparities.

This study comprises a 3-arm parallel cluster randomized controlled trial with low-resourced mothers living in New York City. The study team will randomize fitness class sites (clusters) into Arm A (contact control), receipt of free weekly fitness classes; Arm B, receipt of free childcare combined with free weekly fitness classes; and Arm C, receipt of free childcare combined with free weekly fitness classes and, plus peer support activities. The study team will recruit 90 participants into 3 fitness classes. Physical activity is the primary outcome measured using accelerometers, a self-reported questionnaire, and attendance data. Secondary outcomes (e.g., health status) and mediators/moderators (e.g., social support and cohesion) will be assessed with a baseline and follow-up questionnaire. Ethnographic methods will be used to examine how intersecting forms of social inequality shape women's experiences of physical activity and to understand how real-world conditions shape the intervention implementation. The intention-to-treat analysis will employ linear mixed-effects models (LMM) to assess the main intervention effects on physical activity outcomes and other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Understand/speak English or Spanish
* Have children <12 years old
* Own a mobile phone
* Live in the zip code surrounding as Shape Up NYC sites

Exclusion Criteria:

- Total household income being greater than 165% of the area median income (calculated by household size).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers
Enrollment: 89 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Houghton, PhD, MSc, Principal Investigator — Dept of Epidemiology, MSPH
Locations (3):
- United States (3):
  - Astoria Park, Astoria, New York
  - Crocheron Park, Bayside, New York
  - Forest Park, Richmond Hill, New York

IPD SHARING:
Plan to Share IPD: No
Based on ethical considerations, only the quantitative aggregated data produced in the course of the project will be preserved and shared. The final dataset will include self-reported demographic and behavioral data from surveys and accelerometer data aggregated at the cluster level. To facilitate interpretation of the data, a data dictionary and copies of blank questionnaires will be created, shared, and associated with the relevant datasets.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 89 participants consented but 9 did not complete the baseline assessment, so total 80 participants are counted as part of the study.
Units Other Than Participants: fitness class sites
Groups:
- Enhanced Intervention Arm: Fitness Classes + Childcare + Peer Support: There will be 3 Shape Up NYC classes offered weekly for one hour free of charge to consenting participants in all three arms with a total of 12 classes offered per participant. In addition, they will receive childcare in an adjacent space to the fitness class. In addition to childcare, participants will also receive peer support activities. Peer support activities will consist of group volunteer activities at food pantries, free deliveries of food pantry groceries, and group play dates at local playgrounds. A Community Champion will also facilitate group text messages.
Period: Overall Study
Arm/Group | Control Arm: Fitness Classes Only | Comparator Arm: Fitness Classes + Childcare | Enhanced Intervention Arm: Fitness Classes + Childcare + Peer Support
Started | 26; 1 fitness class sites | 31; 1 fitness class sites | 23; 1 fitness class sites
Completed | 12; 1 fitness class sites | 18; 1 fitness class sites | 8; 1 fitness class sites
Not Completed | 14; 0 fitness class sites | 13; 0 fitness class sites | 15; 0 fitness class sites

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm: Fitness Classes Only | Comparator Arm: Fitness Classes + Childcare | Enhanced Intervention Arm: Fitness Classes + Childcare + Peer Support | Total
Number analyzed (Participants) | 26 | 31 | 23 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 31 | 23 | 80
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 25 | 31 | 23 | 79
  Male | 0 | 0 | 0 | 0
  Unknown/Not reported | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 20 | 17 | 49
  Not Hispanic or Latino | 12 | 11 | 5 | 28
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 5 | 2 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 12 | 12 | 6 | 30
  More than one race | 0 | 4 | 1 | 5
  Unknown or Not Reported | 6 | 10 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 26 | 31 | 23 | 80

OUTCOME MEASURES:

1. Primary Outcome: Total Minutes of Time Spent in Moderate to Vigorous Physical Activity (MVPA)
Description: Weekly MVPA, total physical activity, sedentary time, and sleep will be objectively assessed using a blinded research-grade wrist-worn accelerometer (Axivity AX3) in all groups.
Time Frame: Baseline and follow-up between weeks 10-12
Population: The outcome data are not available for 42 out of the 80 enrolled because participants either did not return their accelerometer or they did not adhere to the protocol of wearing the accelerometer for at least 4 out of the 8 days. 12 unique participants in the Control Arm, 18 unique participants in the Comparator Arm, and 8 unique participants in the Enhanced arm were analyzed for this outcome.
Measure: Least Squares Mean (Standard Error); unit: minutes of MVPA per week
Arm/Group | Control Arm: Fitness Classes Only | Comparator Arm: Fitness Classes + Childcare | Enhanced Intervention Arm: Fitness Classes + Childcare + Peer Support
Number analyzed (Participants) | 12 | 18 | 8
minutes of MVPA per week
  Baseline: number analyzed (Participants) | 8 | 13 | 5
  Baseline | 548 (100.0) | 512 (78.9) | 354 (125.0)
  Follow-up: number analyzed (Participants) | 7 | 11 | 5
  Follow-up | 737 (105.0) | 479 (83.5) | 404 (125.0)

2. Secondary Outcome: EQ5D-5L Score
Description: The EQ5D-5L standardized survey is a generic measure of health status that includes five dimensions: mobility, self-care, usual activities, pain, and anxiety/depression. The EQ-5D-5L index is measured on a total scale from 0 to 1, whereby 0 indicates death and 1 perfect health.
Time Frame: At baseline and follow-up between weeks 10-12
Reporting Status: Not Posted, anticipated posting 2026-04

3. Secondary Outcome: ICEpop CAPability Measure for Adults (ICECAP-A) Score
Description: The ICECAP-A standardized survey captures the broader concept of well-being via five dimensions: feeling settled and secure; love, friendship, and support; being independent; achievement and progress; and enjoyment and pleasure. The ICECAP-A also generates a score between 0 to 1 where one equals 'full capability' and zero equals 'completely incapable'.
Time Frame: At baseline and follow-up between weeks 10-12
Reporting Status: Not Posted, anticipated posting 2026-04

4. Secondary Outcome: Attendance
Description: Shape Up NYC takes attendance at each fitness class, and community champions will take attendance at the peer support activities to understand participation, retention, and attrition levels.
  Attendance rate of all fitness classes will be presented as the mean percent of attendance ([# of participants present in class] divided by [# of available slots] multiplied by 100) over 12 weeks.
Time Frame: 12 weeks
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: Generalized Anxiety Disorder 2-item (GAD-2) Score
Description: The GAD-2 is a brief questionnaire that assesses patient anxiety. The total score range is 0-6, with a higher score indicating worse anxiety.
Time Frame: Baseline and follow-up between weeks 10-12
Reporting Status: Not Posted, anticipated posting 2026-04

6. Secondary Outcome: Patient Health Questionnaire-2 (PHQ-2)
Description: PHQ-2 is a brief questionnaire that assesses frequency of depressed mood and anhedonia. The total score range is 0-6, with a higher score indicating worsening feelings of depression.
Time Frame: Baseline and follow-up between weeks 10-12
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: International Physical Activity Questionnaire (IPAQ) Score
Description: Self-reported physical activity data will be collected using IPAQ. IPAQ asks participants to report the types and frequency of physical activities they have participated in over 7 days. IPAQ score is expressed as median(MET)-min per week: [MET level] x [minutes of activity/day] x [days per week]. It is scored as follows:
  High: Any one of the following two criteria:
  Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week OR 7+ days of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week
  Moderate: Any one of the following three criteria:
  3+ days of vigorous activity, at least 20 minutes per day OR 5+ days of moderate-intensity activity or walking of at least 30 minutes per day OR 5+ days of walking, moderate-intensity or vigorous intensity activities achieving a minimum of 600 MET-min/week.
  Low: Individuals who do not meet criteria for either category
Time Frame: Baseline and follow-up between weeks 10-12
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control Arm: Fitness Classes Only | Comparator Arm: Fitness Classes + Childcare | Enhanced Intervention Arm: Fitness Classes + Childcare + Peer Support
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/31 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/31 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/31 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT06474715/Prot_SAP_000.pdf